CLINICAL TRIAL: NCT00799084
Title: Automated Telephone Monitoring for Symptom Management
Acronym: ATSM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Bill Given, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01CA030724 (NIH)
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Last update posted 2011-12-07 (Estimated); Status verified 2011-12

CONDITIONS: Carcinoma
Keywords: symptom management; cancer; chemotherapy treatment; Behavioral Research; Physiological Effects of Drugs; Clinical Trial, Phase II
MeSH Terms: conditions — Carcinoma; Neoplasms | interventions — Nurses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nurse (Experimental): Receives symptom management assistance from an oncology nurse via the telephone
  Interventions: Behavioral: Nurse
- AVR (Experimental): Receives symptom management assistance from an Automated telephone system
  Interventions: Behavioral: AVR

INTERVENTIONS:
Behavioral: Nurse — Receives 6 telephone calls over 8 weeks from an oncology nurse to assist with symptom management
  Arms: Nurse
Behavioral: AVR — Receives 6 telephone calls over 8 weeks from an programmed automated telephone system to assist with symptom management
  Arms: AVR

SUMMARY:
To improve the management of symptoms, patients with cancer undergoing chemotherapy will be monitored using an automated telephone system to record the severity of 15 prevalent symptoms for up to 8 consecutive weeks. Outcomes include; significant reduction in symptom severity and improvement in health states.

DETAILED DESCRIPTION:
Overview: Prevalent symptoms among patients undergoing chemotherapy include: pain, fatigue, dry mouth, constipation, anorexia, nausea, sleep disturbance, shortness of breath or difficulty breathing, as well as psychological symptoms such as depression and anxiety. A survey of 1000 patients with cancer indicated that close to a quarter reported 10-12 symptoms. Given the impact of symptoms upon physical function, work, emotional distress, and hospitalizations, it is critical that strategies be developed and tested to improve symptom management.

This trial of a behavioural intervention for symptom management is significant because: 1) it contrasts a proactive approach, individualized to patients' symptom management needs, with a more conventional model that places responsibility on the patient for symptom management; 2) it controls for the method of delivery and the use of printed material; 3) it targets prevalent symptoms known to affect cancer patients undergoing chemotherapy; 4) it examines the relative effects of each arm, in terms of symptom severity (primary outcome), impact on patients' physical and social roles, and emotional distress; and 5) it explores these outcomes in terms of their impact on the use of services and costs of care.

Goal: The goal of this randomized trial is to determine if a nurse delivered Patient Assisted Management of Symptoms (PAMS) intervention individualized to patients' needs for symptom management, delivered by telephone, when compared to Telephone Information and Monitoring of Symptoms (TIMS) where symptoms are only monitored by telephone, with references to the symptom management toolkit will reduce symptom severity, improve physical function, and other outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* solid tumor cancer diagnosis
* receiving chemotherapy treatment

Exclusion Criteria:

* Emotional or psychology disorder for which patient is receiving treatment
* does not speak English
* does not have access to a telephone
* difficulty hearing on the telephone

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2003-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Lower reported mean severity index among 7 prevalent symptoms | 9 weeks, 15 weeks

SECONDARY OUTCOMES:
Reduced impact of physical role performance, improved social functioning, and reduced emotional distress; improved levels of communication between patients and providers; and improved patient satisfaction with care. | 9 weeks, 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Charles Given, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States